CLINICAL TRIAL: NCT02492438
Title: Immunogenicity and Safety of the 13-valent Pneumococcal Conjugate Vaccine in Chronic Dialysis Patients That Are 23-valent Pneumococcal Polysaccharide Vaccine Naive and Pre-immunized.
Brief Title: 13 Valent Pneumococcal Conjugate Vaccine in Chronic Dialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AZ Sint-Jan AV (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Vandecasteele Stefaan Johan, Stefaan Johan Vandecasteele, MD, PhD, AZ Sint-Jan AV
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WS2113445
Record Dates: First submitted 2014-08-24; First posted 2015-07-08 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Chronic Kidney Failure
Keywords: pneumococcal vaccination; dialysis; immune response
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PPV23 naive, PPV23 vaccination (Active Comparator): vaccination with PPV-23 in 40 PPV-23 naive patients
  Interventions: Biological: PPV23 vaccination or PCV13 vaccination
- PPV23 naive, PCV13 vaccination (Experimental): vaccination with PCV-13 in 40 PPV-23 naive patients
  Interventions: Biological: PPV23 vaccination or PCV13 vaccination
- PPV23 > 4 years ago, PCV13 vaccination (Experimental): vaccination with PCV-13 in 40 patients that received PPV-23 more than 4 years ago
  Interventions: Biological: PPV23 vaccination or PCV13 vaccination
- PPV23 < 4 years, PCV13 vaccination (Experimental): vaccination with PCV-13 in 40 patients that received PPV-23 less than 4 years ago
  Interventions: Biological: PPV23 vaccination or PCV13 vaccination

INTERVENTIONS:
Biological: PPV23 vaccination or PCV13 vaccination
  Other Names: Prevenar 13; Pneumovac 23

SUMMARY:
To assess the immunogenicity of the PCV13 (13 valent pneumococcal conjugated vaccine) vaccine as compared to the PPV23 (23 valent pneumococcal polysaccharide vaccine) vaccine in patients treated with chronic hemodialysis that are pre-immunized with the PPSV23 vaccine or are PPV23 vaccine naïve by measuring the ELISA and OPA (opsonophagocytic assay) titers after 4 and 52 weeks.

DETAILED DESCRIPTION:
The immunogenicity of the PCV13 (13 valent pneumococcal conjugated vaccine) vaccine as compared to the PPV23 (23 valent pneumococcal polysaccharide vaccine) vaccine in patients treated with chronic hemodialysis that are pre-immunized with the PPV23 vaccine or are PPV23 vaccine naïve will be measured by ELISA and OPA (opsonophagocytic assay) titers after 4 and 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. they are under chronic dialysis treatment
2. are 50 years or older and not pregnant
3. have no immediate life threatening conditions
4. are not allergic to one of the compounds of the vaccine
5. have a known pneumococcal vaccination status
6. give their informed consent.

Exclusion Criteria:

Patients not fulfilling the inclusion criteria.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2013-02; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Antibody response after vaccination to involved serotypes measured by OPA and ELISA | 52 weeks after vaccination

SECONDARY OUTCOMES:
record of side effects of vaccination | first week after vaccination
Antibody response after vaccination to involved serotypes measured by OPA and ELISA | 4 weeks after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Stefaan J Vandecasteele, MD, PhD, Principal Investigator — Department of Nephrology and Infectious Diseases, AZ Sint-Jan Brugge, Belgium
Locations (2):
- Belgium (2):
  - Dienst Nefrologie, OLV Ziekenhuis, Aalst
  - AZ Sint-Jan Brugge Oostende AV, Bruges